CLINICAL TRIAL: NCT00846352
Title: Randomized Trial Comparing Early Versus Late Bronchoscopy in Hematopoietic Stem Cell Transplant Patients With Pulmonary Infiltrates.
Brief Title: Early Versus Late Bronchoscopy in Bone Marrow Transplantation (BMT) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Ohio State University (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00007668
Record Dates: First submitted 2009-02-02; First posted 2009-02-18 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2009-08

CONDITIONS: Bone Marrow Transplantation
Keywords: Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation; Bronchoscopy
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Bronch (Active Comparator): This group will receive bronchoscopy within 36 hours of enrollment into the study.
  Interventions: Procedure: Variation in the time for performing bronchoscopy
- Late bronch (Active Comparator): This group will receive bronchoscopy within 5 days of enrollment.
  Interventions: Procedure: Variation in the time for performing bronchoscopy

INTERVENTIONS:
Procedure: Variation in the time for performing bronchoscopy — The study will compare outcomes amongst patients assigned to receive early bronchoscopy (within 36 hours of enrollment)versus those in whom bronchoscopy is delayed (5 days after enrollment).
  Other Names: Bronchoscopy

SUMMARY:
This study will evaluate the outcomes of bronchoscopy in Bome Marrow Transplant (BMT) patients who develop lung infiltrates suspicious for infections of the lungs. It will consist of two groups, one group will receive bronchoscopy within thirty six hours of enrollment, while the other group will receive bronchoscopy five days after enrollment. The purpose of this study is to determine the ideal time for bronchoscopy in this group of patients.

DETAILED DESCRIPTION:
At this time there exist no studies that help Pulmonologists and Oncologists decide on the best time to perform diagnostic bronchoscopies in Bone Marrow Transplant patients with suspected pulmonary infections. Practice patterns vary from institution to institution and also vary widely within an institution based on the practice preferences of the attending physicians. This study is a prospective randomized trial comparing early ( within 24-36 hours of enrollment) to late ( day 5-6 after enrollment) bronchoscopy in Bone Marrow Transplant patients who develop pulmonary infiltrates or clinical evidence of respiratory infection. If patients in the late arm require earlier bronchoscopy or do not require bronchoscopy on day 5-6 then the care will be dictated by the attending physician. Only bronchoscopies that are clinically indicated will be performed.

The aim is to determine the optimal timing for performing bronchoscopy in this group of patients. The primary outcomes will be change of therapy as determined by addition or removal of antibiotics, antifungals, antivirals or steroids etc. as well as the oncologist's opinion on the impact the bronchoscopic results had on care of the patient. Patients will be followed throughout their hospitalization as well as receive a phone call 3 months after hospital discharge. Written consent will be obtained from the patients or health care power of attorney in relevant cases.

It is our hope that the results of this study will help better define the role of bronchoscopy in the management of Bone Marrow Transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had allogenic or autologous HSCT who are admitted to the BMT, and felt to need bronchoscopy by their physician.

Exclusion Criteria:

* Active hemoptysis, allergies to topical and IV anesthetics with no appropriate substitutes available. Being on non-invasive positive pressure ventilation that would not allow for safe bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-08-02 (Actual); Study Completion 2010-08-02 (Actual)

PRIMARY OUTCOMES:
Change in therapy due to results obtained from bronchoscopy. | When results of bronchoscopy are available

SECONDARY OUTCOMES:
In-Hospital and three month mortality | Three months from time of enrollment
Duration of antibiotic therapy | Variable

CONTACTS AND LOCATIONS:
Overall Officials: John F Conforti, D.O, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - The University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Kantrow SP, Hackman RC, Boeckh M, Myerson D, Crawford SW. Idiopathic pneumonia syndrome: changing spectrum of lung injury after marrow transplantation. Transplantation. 1997 Apr 27;63(8):1079-86. doi: 10.1097/00007890-199704270-00006. PMID 9133468
- [Background] Krowka MJ, Rosenow EC 3rd, Hoagland HC. Pulmonary complications of bone marrow transplantation. Chest. 1985 Feb;87(2):237-46. doi: 10.1378/chest.87.2.237. PMID 2981658
- [Background] Seiden MV, Elias A, Ayash L, Hunt M, Eder JP, Schnipper LE, Frei E 3rd, Antman KH. Pulmonary toxicity associated with high dose chemotherapy in the treatment of solid tumors with autologous marrow transplant: an analysis of four chemotherapy regimens. Bone Marrow Transplant. 1992 Jul;10(1):57-63. PMID 1515880
- [Background] Rano A, Agusti C, Jimenez P, Angrill J, Benito N, Danes C, Gonzalez J, Rovira M, Pumarola T, Moreno A, Torres A. Pulmonary infiltrates in non-HIV immunocompromised patients: a diagnostic approach using non-invasive and bronchoscopic procedures. Thorax. 2001 May;56(5):379-87. doi: 10.1136/thorax.56.5.379. PMID 11312407
- [Background] White P, Bonacum JT, Miller CB. Utility of fiberoptic bronchoscopy in bone marrow transplant patients. Bone Marrow Transplant. 1997 Oct;20(8):681-7. doi: 10.1038/sj.bmt.1700957. PMID 9383232